CLINICAL TRIAL: NCT06226753
Title: Impact of General Anesthesia v/s Spinal Anesthesia on Enhanced Recovery After Surgery (ERAS) Parameters in Intestinal Stoma Reversal: A Randomised Control Trial
Brief Title: Impact of General Anesthesia v/s Spinal Anesthesia on ERAS Parameters in Intestinal Stoma Reversal
Acronym: SPIGERAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Tushar Subhadarshan Mishra, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG Thesis/2023-24/81
Record Dates: First submitted 2024-01-03; First posted 2024-01-26 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; ERAS; Surgical Stomas; Ileostomy - Stoma; Colostomy Stoma

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized. Intervention Model: Open labeled, Parallel Assignment, Superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stoma reversal under GA (Active Comparator): Loop ileostomy closure will be performed under General anaesthesia
  Interventions: Procedure: Type of anaesthesia used
- Stoma reversal under SA (Experimental): Loop ileostomy closure will be performed under Spinal anaesthesia
  Interventions: Procedure: Type of anaesthesia used

INTERVENTIONS:
Procedure: Type of anaesthesia used — Spinal anaesthesia will be used for closure of loop ileostomy
  Other Names: ERAS

SUMMARY:
Randomized, Interventional ,Open labeled, Parallel Assignment and Superiority trial.

DETAILED DESCRIPTION:
Temporary intestinal stomas are commonly created in emergency and elective surgeries to divert intestinal contents from distal anastomoses site or after resection of a diseased bowel segment. They however increase the morbidity of a patient, impacting the life of a patient socially and psychologically. A timely and planned early stoma reversal can reduce various stoma related complications (up to 71%) like parastomal leakage, dermatitis, prolapse, retraction, dehydration, electrolyte imbalance and acute kidney injury, and occasionally requirement of parenteral nutrition. However these patients are often subject to long waiting periods for want of availability of a slot under general anaesthesia. More importantly, quite some of these patients with temporary stoma have poor general condition and comorbidity prohibiting a timely stoma closure. Closing intestinal stomas under regional anaesthesia could have partially addressed the issue. But studies exploring the feasibility of the stoma closure under spinal/ regional anaesthesia are limited to a few case series. There is a dearth of good quality literature having a head to head comparison ileostomy closure done under spinal anaesthesia vs those done under the more commonly employed general anaesthesia. ERAS was brought into picture considering the physiological changes in metabolism during the perioperative period and implemented to cut short the phase of perioperative stress and early recovery of the patient, with minimal postoperative complications ERAS is an evidence based multidisciplinary approach that has outweighed many conventional approaches to achieve early discharge of the patient in various elective and emergency surgeries like Colorectal, Gastric, Hepatobiliary, Breast and Pre pyloric perforation Dr Henrik Kehlet, a Danish Colorectal Surgeon first proposed the concept of Fast track surgery in order to decrease the surgical stress, the different components being broadly classified into Preoperative, intra-operative and post-operative care. ERAS can potentially be implemented in Intestinal Stoma Reversal Surgery, and is worth demanding of a Day Care Surgery, with Spinal Anaesthesia expecting to be an adjunct in fastening the recovery.

Preoperative Preoperative counselling Avoid prolong fasting Carbohydrate loading No preanaesthetic medication Antibiotic prophylaxis Thromboprophylaxis

Intraoperative Short acting anaesthetics. Minimaly invasive surgery Goal directed fluid therapy Temperature homeostasis

Postoperative Prevention of PONV Early removal of catheter and drain. Early enteral nutrition Early mobilization

STUDY OBJECTIVES PRIMARY OBJECTIVE To study the return of bowel function Secondary Objective Return of functional parameters Complication rates Post operative pain assessment Surgeon and patient comfort

RATIONALE Feasibility of intestinal stoma closure has the potential to avoid general anaesthesia and its related delays in the recovery. Stoma Reversal under Spinal Anaesthesia if found to be feasible, will be less taxing on the waiting list under GA and will achieve better perioperative course compared to GA.

NOVELTY July 2005 saw the publication of a case series demonstrating the effectiveness of Spinal Anaesthesia for stoma reversal in a high-risk patient. [8] However, there is no RCT or any other reasonable quality study that compares outcome of stoma reversal with SA v/s GA. This will also be the first study comparing the effect of Spinal anaesthesia v/s GA on the different parameters of ERAS guidelines.

HYPOTHESIS In a study on LSCS, spinal anaesthesia showed earlier return of bowel function. [9] So we hypothesise that spinal anaesthesia will lead to earlier return of functional parameters in stoma closure too.

REVIEW OF LITERATURE KEYWORDS 'Loop ileostomy', 'stoma', 'stoma reversal', 'stoma closure', 'Spinal Anaesthesia' , '', 'ERAS',' local anesthesia','fastrack surgery' SEARCH GOAL To find literature which studies the efficacy of spinal anaesthesia in stoma reversal (or other Gastrointestinal Surgeries) and its impact on the hospital stay of patients.

Also studies that implemented certain measures which led to early recovery in such patients were looked for.

STRATEGY Searches were made in following databases: PubMed, Google Scholar Search terms included 'Loop ileostomy', 'stoma', 'stoma reversal', 'stoma closure', 'Spinal Anaesthesia', 'ERAS',' local anesthesia','fastrack surgery' A case series of 6 patients under high risk revealed reversal of loop ileostomy can be performed safely and comfortably under spinal anaesthesia Favourable outcomes were -patients were able to resume normal oral diet in the immediate post-operative period, and on POD 2 patient were discharged A prospective study comparing overall outcome under GA v/s SA in LSCS showed earlier return of functions in SA over GA, paving way for incorporating ERAS into this study.

MATERIALS AND METHODS STUDY SETTING: Patients undergoing Stoma Reversal at All India Institute of Medical Institute, Bhubaneswar in the Department of General Surgery, Department of Surgical Gastroenterology, Surgical Oncology and Department of Anaesthesia STUDY TYPE: Interventional. STUDY DESIGN: Allocation: Randomized. Intervention Model: Open labeled, Parallel Assignment, Superiority trial. Primary Purpose: Treatment. RANDOMIZATION: Simple randomization, Allocation concealment: Serially Numbered Opaque Sealed Envelope technique Point of randomization: Preoperative after fitness for stoma reversal.

SAMPLE SIZE Sample Size Calculation

The sample size for the study was based on (Havas et al, 2013), who reported the mean time to passage of flatus in the two groups as follows:

Parameter Group 1: Mean ± SD Group 2: Mean ± SD 19±17.8 24±16

The sample size required in each arm of the study was calculated according to the formula given by Snedecor & Cochran (1989):

Sample size (N) = 1 + 2(Zα + Z1-β)¬2 σ2 δ2

Where:

σ (Pooled SD) = 16.9 δ (Difference of Means) = 5. However, we calculated a sample size to detect a difference as low as 12 hours Type I error (α) = 5%, Zα (Value of Standard Normal Distribution for α = 5%) = 1.96 Type II error (β) = 10%, Power (1 - β) = 90%, Z1-β = 1.282

Based on the formula given above, using the mentioned values, the sample size required is:

Sample size (N) = 1 + 2(1.96 + 1.282)¬2 16.92 122 = 42.8 ≈ 43 Allowing for 10% attrition, we get a sample size of 43/0.9 ≈ 50 Thus, assuming 90% Power and 95% Confidence interval, the minimum calculated sample size for each arm is 50 (total = 100).

METHODS USED The parameters that will be compared will be the safety (leaks), feasibility (intraoperative pain in spinal arm, conversions to GA) and quality of life at 6 hours and 24 hours in the perioperative period. Requirement of analgesia after the perioperative analgesics given in the OT will be recorded in. ERAS guidelines will be followed in either arm and the impact of each type of anaesthesia over the protocol will be studied. The return of functional parameters will be recorded and compared in either arm Preoperative

* Routine management as advised in PAC.
* Bowel wash preparation would be done.
* Counselling of patient
* Nasogastric tube aspiration
* Intravenous fluids Intra-operative
* Bowel anastomosis of Loop, Double barrel or End stoma with hitched distal loop to be done either with hand sewn or stapler method ERAS Anesthesia protocol [12]
* Near zero fluid balance at 1-3 ml/kg/hour. Low threshold to begin Noradrenaline to keep -MAP>60mmHg
* Short acting anesthetic agents and short acting muscle relaxants
* Intraoperative warming Group A GA- General Anesthesia with Tracheal Intubation+ TAP block Low tidal volume ventilation Group B SA-
* SA with 10 to 15 mg of Hyperbaric Bupivacaine and 25 mcg of Fentanyl
* If case of pain, top up with Local anesthesia (0.5% Lignocaine with Adrenaline) will be infiltrated. The number of times this would be required be recorded for analysis.
* Using a parastomal incision
* NG tube and Foley's removed on table after surgery Post-operative
* Inj PCM 1g iv QID will be given for first 24 hrs
* After 24 Hr oral analgesics Tab Paracetamol 650 mg QID will be used.
* Analgesia on demand - Rescue analgesic (Inj. Tramadol 100 mg iv ) will be used if NRS > 4 or if patient demands and the total dose recorded.
* Oral clear liquid sips will be given after 4 hours and oral unrestricted clear liquids after 12 hours in both the arms
* IV fluid will be discontinued as soon as the patient takes sufficient liquids semi solids to compensate for the daily calories requirement of the body.
* Early ambulation within 2 hours in either arm.
* NG Tube will be re-inserted in patients developing vomiting and signs of paralytic ileus and tube will be removed once vomiting subsides
* Foley's catheter will be re inserted in patients developing urinary retention and will be removed once retention subsides CRITERIA FOR DISCHARGE ( All criteria to be fulfilled)
* Adequate pain relief on oral analgesia (patients not needing injectable for more than 12 hours)
* Accepting at least oral semisolid diet with no PONV or distension of abdomen and is off IV fluids
* Able to ambulate without support as per criteria for discharge after regional anaesthesia as a Day Case Surgery- normal perianal sensation (S4-S5), ability to plantar reflex the foot and proprioception of great toe.[13]

STATISTICAL ANALYSIS PLAN Data will be entered in Microsoft excel, and analysis will be done using the latest version of IBM SPSS software.

ETHICAL ISSUES

* Approval shall be taken from the Ethics Committee of the All India Institute of Medical Sciences, Bhubaneswar.
* Informed written consent will be obtained from patient/patient attenders in their own understandable language.
* A participant information sheet will be provided to the patients.
* Participants will be explained that their identity will remain confidential.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient ;18 years
* Patients with Loop stoma, Double Barrel Stoma or End stoma with
* documented hitched distal loop.
* Patients evaluated and fit for surgery

Exclusion Criteria:

* Patients requiring mid line laparotomy for stoma reversal
* Patient having active stoma related complications like high output stoma
* and dehydration - Acute Kidney Injury, stoma prolapse, etc making them
* unfit for surgery.
* Patient denying consent for SA or ERAS protocol
* Patient having contraindication for either type of anaesthesia (where
* randomisation would not be possible)
* Patient needing to be converted to GA after pain /discomfort experienced
* by patient or if there was failed spinal anaesthesia
* Patient having abnormal coagulation profile
* Coexistent neurological or psychiatric illness or unable to understand the
* study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time to passage of flatus | Up to 72 hours after surgery
  Time to passage of first flatus from the time of patient leaving operating room up to 72 hours after surgery will be estimated in hours

SECONDARY OUTCOMES:
Time to passage of motions | Up to 1 week after surgery
  Time to passage of first stool from the time of patient leaving operating room up to 1 week after surgery in hours will be estimated
Time taken to resumption of oral intake | Up to 72 hours after surgery
  Time to resume the first oral intake from the time of patient leaving operating room up to 72 hours after surgery will be estimated in hours
Time of complete stoppage of IV fluids | Up to 72 hours after surgery
  Time to completely stop the administration of intravenous fluids from the time of patient leaving operating room up to 72 hours after surgery will be estimated in hours

OTHER OUTCOMES:
Postoperative mean Numerical Rating Score | At 6,12 and 24 hours
  Postoperative pain score will be estimated. Numerical Rating Score will be used- Minimum 0 and Maximum 10
Time to need 1st injectable rescue analgesic i.e. Tramadol | Up to 72 hours after surgery
  Time of requirement of rescue analgesics from the time of patient leaving operating room up to 72 hours after surgery will be estimated in hours
Total number of doses of rescue analgesic used | Up to 1 week after surgery
  Total number of doses of rescue analgesics used from the time of patient leaving operating room up to 1 week after surgery will be calculated
Surgeon's and patient satisfaction by Local Experienced Discomfort Score | Intraoperative, From the time of incision to time of completion of skin closure
  Degree of satisfaction of the surgeon and the patient for the procedure performed from the time of incision to time of completion of skin closure will be noted. Local Experienced Discomfort Score will be used- Minimum 0 and Maximum 10
Percentage of times there is a need of conversion of Spinal Anesthesia to General Anesthesia intraoperative pain or severe discomfort to the patient | Intraoperative, From the time of patient entering operating room to leaving operating room
  Number of times there was need to administer General anesthesia in procedures under spinal anesthesia
Percentage of times there is a need for ICU admission for anesthesia recovery related issues | Immediately after the intervention, Up to 24 hours after surgery
  Number of times postoperative ICU stay from the time of patient leaving operating room up to 24 hours after surgery
Duration of post-operative hospital stay | Immediately after the intervention
  Length of hospital stay from the time of patient leaving operating room up to discharge
Complications and its incidence: ileus, need for RT insertion or readmission, anastomotic leak ( in terms of Clavein Dindo Classification) | Postoperative, Upto 30 days from surgery
  Any complication after surgery will be noted
Time to walk around independently | Up to 72 hours after surgery
  Time to start ambulation from the time of patient leaving operating room up to 72 hours after surgery will be noted in hours
Duration of Surgery | From the time of incision to time of completion of skin closure
  Duration of Surgery from the time of incision to time of completion of skin closure will be noted in hours
Duration of Stay in Operating Room | From the time of patient entering operating room to leaving operating room
  Duration of Stay in Operating Room from the time of patient entering operating room to leaving operating room will be recorded in hours

CONTACTS AND LOCATIONS:
Overall Officials: Tushar S Mishra, MBBS MS, Principal Investigator — AIIMS Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences,, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No